CLINICAL TRIAL: NCT01320813
Title: Randomized Trial Comparing Complication Rates Associated With Robot-assisted Thyroidectomy to External Thyroidectomy
Brief Title: Trial Comparing Complication Rates Associated With Robot-assisted Thyroidectomy to External Thyroidectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find enough patients who accept randomization of surgical procedures.
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC-I/2010/BL-01; 2011-A00049-32 (Other: RCB number)
Record Dates: First submitted 2011-03-22; First posted 2011-03-23 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Thyroid Nodule; Goiter; Thyroiditis; Graves Disease
Keywords: da vinci robot; Thyroidectomy
MeSH Terms: conditions — Thyroid Nodule; Goiter; Thyroiditis; Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Robot arm (Experimental): Patients in this arm will have a thyroidectomy performed using a robot-assisted endoscopic technique.
  Interventions: Procedure: Robot-assisted thyroidectomy
- Open surgery (Active Comparator): Patients in this arm will have a thyroidectomy using an open surgical technique.
  Interventions: Procedure: Open thyroidectomy

INTERVENTIONS:
Procedure: Robot-assisted thyroidectomy — Patients will have a thyroidectomy via a robot-assisted (da Vinci robot) endoscopic (subclavical entry)surgical technique.
  Arms: Robot arm
Procedure: Open thyroidectomy — Patients will have a conventional (non-endoscopic) thyroidectomy using an open surgical technique
  Arms: Open surgery

SUMMARY:
The main objective is to compare 12 month complication rates between a new surgical method for thyroidectomy (robot-assisted endoscopic thyroidectomy via a sub-clavical approach) and open thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 12 months of follow-up
* The patient is a candidate for total thyroidectomy because of a nodular pathology, a diffuse goiter, thyroiditis, or Basedow's disease
* Patient has calcitoninemia < 9 ng/pl
* Patient has normal calcemia
* Patient has PTH level between 5 ng/l and 75 ng/l
* The subject has a normal laryngeal mobility

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* The patient is pregnant
* The patient is breastfeeding
* The patient is not available for 12 months of follow-up
* Subject has a preoperative diagnosis of cancer on fine needle aspiration biopsy of the thyroid or cervical lymph node
* Lymph node metastasis strongly suspected clinically and/or sonographically
* The subject has an extension of substernal thyroid (diving goiter)
* Family history of medullary thyroid cancer
* The subject has a history of neck surgery
* Contraindication for general anesthesia

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Presence/absence of complications (composite score) | 12 months
  The per or post-operative occurrence of at least one of the following: postoperative hemorrhage requiring reintervention; cervical infection requiring antibiotics and/or surgical intervention; transient or persistent laryngeal paralysis; transient or persistent hypoparathyroidy (calcemia < 1.9 µmol/l). Transiient means < than and persistent means >= 12 months.

SECONDARY OUTCOMES:
Incision size (mm) | 12 months
  Length of incision in the open group, and sum of incision lengths in the robot group.
Patient satisfaction score | 12 months
  Patient satisfaction as regards the incision scar measured using a visual analog scale from 0.0 to 10.0.
Presence/absence of conversion to open technique | 1 day
  For patients in the robot arm: presence/absence of conversion to open technique.
Operating room prep time (min) | 1 day
  Time in minutes necessary to prep the operating room
Presence/absence of per-operative complications | 1 day
  Presence/absence of per-operative complications
Hospital stay (d) | 7 to 15 days post-op
  Length of hospitalization in days required after thyroidectomy
Change in thyroglobulinemia (ng/l) | 12 months
  Thyroglobulinemia at 12 months - Thryoglobulinemia as baseline
Change in calcemia (mg/l) | Day 1
  Calcemia on Day 1 - Calcemia at inclusion
Change in calcemia (mg/l) | Day 7 to 15
  Calcemia at the control visit (days 7 to 15) - Calcemia at inclusion
Change in calcemia (mg/l) | 12 months
  Calcemia at 12 months - Calcemia at inclusion
Change in phosphoremia (mg/l) | Day 1
  Phosphoremia at 1 day postop - Phosphoremia at inclusion
Change in phosphoremia (mg/l) | Days 7 to 15
  Phosphoremia at control visit (days 7 to 15) - Phosphoremia at inclusion
Change in phosphoremia (mg/l) | 12 months
  Phosphoremia at 12 months - Phosphoremia at inclusion
Change in parathormonemia (ng/l) | Day 1
  Parathormonemia on Day 1 post-op - parathormonemia at inclusion
Change in parathormonemia (ng/l) | Days 7 to 15
  Parathormonemia at control visit (days 7 to 15) - parathormonemia at inclusion
Change in parathormonemia (ng/l) | 12 months
  Parathormonemia at 12 months - parathormonemia at inclusion
Visual Analog Pain Score | Day 1
  Visual Analog Scale for pain (0.0 to 10.0)
Visual Analog Pain Score | Days 7 to 15
  Visual Analog Scale for pain (0.0 to 10.0)
Visual Analog Pain Score | 12 months
  Visual Analog Scale for pain (0.0 to 10.0)
Direct medical costs (€) | 12 months
Indirect medical costs (€) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Lallemant, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard, France